CLINICAL TRIAL: NCT01864096
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Metformin in Reducing Progression Among Men on Expectant Management for Low Risk Prostate Cancer: The MAST (Metformin Active Surveillance Trial) Study
Brief Title: The Metformin Active Surveillance Trial (MAST) Study
Acronym: MAST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAST 01
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Prostate Cancer
Keywords: localized; prostate; cancer; metformin; active surveillance
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin 850 mg, twice daily for 36 months
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo tablets, 2teice daily for 36 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — One month run-in of 850mg metformin once daily, followed by 850mg twice daily of metformin for 35 months. Total time is 36 months.
  Other Names: Metformin hydrochloride
  Arms: Metformin
Drug: Placebo — One month run-in of placebo tablet once daily, followed by twice daily for 35 months. Total time is 36 months.
  Other Names: Placebo tablet
  Arms: Placebo

SUMMARY:
This study aims to see if metformin can delay the time to progression in men with low risk prostate cancer when compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Must be male > 18 and < 80 years of age
2. Have biopsy proven, low-risk, localized prostate cancer choosing expectant management as primary treatment ≤ 1year. [For the purposes of assessing subject eligibility a diagnostic biopsy must have included at least 10 cores, ≤1/3 of total number of cores sampled and < 50% of any one core positive) and must have been obtained within 6 months of screening]. Initial diagnosis of T1a/T1b obtained during a TURP is not allowed
3. Gleason score ≤ 6 [Gleason pattern 4 or above must not be present on any biopsy (initial or entry)]
4. Clinical stage T1c-T2a
5. Serum PSA ≤10 ng/mL (prior to biopsy)
6. Life expectancy greater than 5 years, as judged by the treating clinician/urologist
7. Able to swallow and retain oral medication
8. Hemoglobin A1c < 6.5%
9. Able and willing to participate in the full 3 years of the study
10. Able to understand instructions related to study procedures
11. Able to read and write (health outcome questionnaires are self-administered), understand instructions related to study procedures and give written informed consent

Exclusion Criteria:

1. Subject that has ever been treated for prostate cancer with any of the following:

   * Radiotherapy (external beam or brachytherapy)
   * Chemotherapy
   * Hormonal therapy (e.g., megestrol, medoxyprogesterone, cyproterone)
   * Oral glucocorticoids
   * GnRH analogues (e.g., leuprolide, goserelin, degarelix)
2. Current and/or previous use of the following medications:

   * Use of 5α-reductase inhibitors (eg. Finasteride, Dutasteride) within the past 6 months of screening
   * Drugs with antiandrogenic properties (e.g., flutamide, bicalutamide, ketoconazole, progestational agents) within 6 months prior to screening
3. Previous or current diagnosis of type 1 or type 2 diabetes
4. Exposure to metformin within 12 months of screening
5. Planned or concurrent use of metformin hydrochloride, sulfonylureas, thiazolidinediones, or insulin for any reason
6. Known hypersensitivity or intolerance to metformin hydrochloride
7. Any condition associated with increased risk of metformin hydrochloride-associated lactic acidosis (e.g. congestive heart failure defines as NYHA class III or IV, history of any type of acidosis, habitual intake of ≥ 4 alcoholic beverages per day)
8. Subject has had prior prostatic surgery including TUNA, TURP, TUIP, laser treatment, thermotherapy, balloon dilatation, prosthesis, and ultrasound ablation within 3 months of screening
9. Participation in any investigational or marketed drug trial within 30 days prior to screening or anytime during the study period. This includes any interventional or exercise trials
10. Any unstable serious co-existing medical condition(s) including, but not limited to, myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to Screening visit
11. Abnormal liver function test:

    * Total bilirubin > 1.8 X institutional upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) > 1.8 X institutional ULN
    * Alanine aminotransferase (ALT) > 1.8 X institutional ULN
    * Alkaline phosphatase (ALP) > 1.8 X institutional ULN
12. Serum creatinine > 1.8 X ULN
13. History of other malignancies, with the exception of adequately treated nonmelanoma skin cancer, stage I melanoma, NMIBC or other solid tumors curatively treated with no evidence of disease for at least 5 years
14. History or current evidence of substance abuse, as defined in DSM-IV, within 12 months of screening
15. History of any illness (including psychiatric) that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject
16. No other concurrent metformin hydrochloride, sulfonylureas, thiazolidinediones, or insulin for any reason

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2013-10; Primary Completion 2024-02-16 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Time to progression | 3 years
  Time to progression - progression is defined as the earliest of the following events:
  1. Primary therapy for prostate cancer (e.g. prostatectomy, radiation, hormonal therapy)
  2. Pathological progression as defined as one of the following:
  i. >1/3 of total amount of cores involved ii. At least 50% of any one core involved iii. Gleason pattern 4 or higher

SECONDARY OUTCOMES:
Time to primary therapy for prostate cancer | 3 years
  Length of time before the participants move on to more radical treatment options (prostatectomy, radiation and/or hormonal therapy)
Time to pathological progression | 3 years
Change from baseline in disease-related patient anxiety | 3 years
  Measured by the Memorial Anxiety Scale for Prostate Cancer (MAX-PC)
Change from baseline in decisional satisfaction and decisional conflict | 3 years
  Measured by the Decisional Regret scale
Change from baseline in prostate cancer diagnosis at repeat biopsy | 3 years
Change in Gleason Score at repeat biopsy | 3 years
Change in clinical stage of prostate cancer based on digital rectal examination | 3 years
Assess the prognostic and predictive value of prostate cancer biomarkers | 3 years
  Using biomarkers in tissue, blood and urine samples
To determine the safety and incidence of (serious) adverse events from the administration of 36 months of metformin to men with early stage prostate cancer | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Neil Fleshner, MD, MPH, FRCSC, Principal Investigator — University Health Network: Department of Surgical Oncology (Urology); Anthony Joshua, MD, Principal Investigator — University Health Network: Department of Surgical Oncology (Urology)
Locations (12):
- Canada (12):
  - Manitoba Cancer Care Centre, Winnipeg, Manitoba
  - CDHA - Victoria Site, Halifax, Nova Scotia
  - McMaster Institute of Urology-St .Joseph's Healthcare, Hamilton, Ontario
  - Centre for Appled Urologic Research, Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre-Victoria Hospital, London, Ontario
  - Ottawa Hospital Research Institute (The Ottawa Hospital), Ottawa, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre L'Hopitalie de l'Universite de Montreal, Montreal, Quebec
  - MUHC - Montreal General Hospital, Montreal, Quebec
  - Centre de Recherche du CHUS, Sherbrooke, Quebec
  - Alberta Urology Institute, Edmonton